CLINICAL TRIAL: NCT00724906
Title: Evaluation of the Diagnostic Accuracy and Safety of 123 I-ALTROPANE® as an Imaging Agent to Aid in the Diagnosis of Parkinsonian Syndromes (POET-2)
Brief Title: Two Separate But Identical Studies Evaluating the Safety and Efficacy of ALTROPANE® in the Use of SPECT Imaging for Upper Extremity Tremor
Acronym: POET-2
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Alseres Pharmaceuticals, Inc (Industry)
Responsible Party: Susan M. Flint, M.S., R.A.C., C.C.R.A., C.C.R.P. Senior VP Drug Development, Alseres Pharmaceuticals, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ALSE-A-02a, ALSE-A-02b
Record Dates: First submitted 2008-07-28; First posted 2008-07-30 (Estimated); Last update posted 2010-02-03 (Estimated); Status verified 2010-02

CONDITIONS: Parkinsonian Syndromes
Keywords: Essential Tremor; Parkinsonian Tremor; Parkinson Disease; Upper Extremity Tremor with duration of less than 2 years; Diagnosis; Subjects; Upper; Extremity; Tremor; Less; Than 2 years
MeSH Terms: conditions — Parkinsonian Disorders; Essential Tremor; Parkinson Disease; Disease; Tremor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Parkinsonian Syndromes (Experimental): Subjects with Parkinsonian Syndromes
  Interventions: Drug: 123 I - ALTROPANE®
- Non-Parkinsonian Syndromes (Experimental): Subjects with Non-Parkinsonian Syndromes
  Interventions: Drug: 123 I - ALTROPANE®

INTERVENTIONS:
Drug: 123 I - ALTROPANE® — 8.0 mCi (±1.0 mCi) will be administered intravenously to each subject.

SUMMARY:
This will be two separate but identical studies: ALSE-A-02a, ALSE-A02b. Each study is designed to evaluate the diagnostic accuracy and safety of a single dose of 123I-ALTROPANE® in subjects with upper extremity tremor for less than three years. Currently, no radiopharmaceutical diagnostic imaging agent has been approved by the FDA in the U.S. for use in diagnosing Parkinson disease and related Parkinsonian syndromes. The diagnosis of Parkinsonian syndromes in the U.S. is based on clinical criteria only. The goal is to demonstrate that 123I-ALTROPANE® paired with SPECT imaging permits a more accurate early diagnosis of Parkinson disease than a clinical diagnosis by a general neurologist.

DETAILED DESCRIPTION:
Each study is a prospective, multi-center, non-randomized, open-label, out patient clinical trial which will include up to 240 subjects per study. Subjects will be male and female, age 40-80 years, with approximately 20 sites per study.

Subjects will participate in 5 study visits over the course of the study period. The screening visit will include an assessment of eligibility. The second visit will be the collection of the community neurologist's diagnostic assessment. The third visit, during which all subjects receive a single intravenous (IV) injection of 123I-ALTROPANE® and single photon emission computed tomography (SPECT) imaging, will include appropriate safety assessments before and after dosing. The fourth visit, to occur 24 to 72 hours after SPECT imaging, will include follow up safety assessments as well as the first Movement Disorder Specialist's (MDS) evaluation. The fifth visit, to occur 6 months (±7 days) after SPECT imaging, will include follow-up safety assessments as well as the MDS reevaluation and truth standard diagnosis. The subject's participation in the study will be up to 7 months.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must provide written informed consent prior to the initiation of any study related procedures;
2. Age 40 to 80 years;
3. Subjects must have had upper extremity tremor for < 3 years duration.

Exclusion Criteria:

1. Any clinically significant acute or unstable physical or psychological illness based on medical history or physical examination at Visit 1, as determined by the PI;
2. Any unexpected clinically significant abnormal laboratory or electrocardiogram (ECG) results obtained at Visit 1 and as determined by the PI;
3. Any history or drug, narcotic, or alcohol abuse within 2 years before the date of informed consent, as defined by the Diagnostic and Statistical Manual of the American Psychiatric Association, Fourth Edition, revised DSM-IVR, American Psychiatric Association, 1994;
4. Positive drug screen for opiates, cocaine or amphetamines at Visit 1;
5. Positive pregnancy test at Visit 1 and/or Visit 3;
6. Participation in an investigational drug or device clinical trial within 30 days prior to the date of informed consent;
7. Previous participation in any 123I-ALTROPANE® trial;
8. Any exposure to radiopharmaceuticals within 30 days prior to the date of informed consent;
9. Breast-feeding;
10. Inability to lie supine for 1 hour;
11. Any thyroid disease other than treated hypothyroidism;
12. Known sensitivity or allergy to iodine or iodine containing products;
13. Treatment within the 4 weeks before the date of the informed consent with buproprion, methylphenidate or amphetamine;
14. Any treatment with anti-Parkinson's drugs within 4 weeks before the date of informed consent.

Subject eligibility based on exclusion criteria 1, 2, 3, 4, and 20 will be confirmed at Visit 3 prior to dosing.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2010-07; Primary Completion 2011-07 (Estimated); Study Completion 2011-07 (Estimated)

PRIMARY OUTCOMES:
To evaluate the diagnostic accuracy of a single dose of 123 I-ALTROPANE® as an imaging agent to aid in the diagnosis of Parkinsonian syndromes (PS) in subjects with upper extremity tremor for less than 2 years. | 7 months

SECONDARY OUTCOMES:
To evaluate the safety of 123 I-ALTROPANE® in subjects with upper extremity tremor for less than 2 years. | 7 months

CONTACTS AND LOCATIONS:
Locations (1):
- Alseres Pharmaceuticals, Inc, Hopkinton, Massachusetts, United States